CLINICAL TRIAL: NCT07324005
Title: Efficacy of Combining Ultrasound-Guided Needle Release of Transverse Carpal Ligament and Median Nerve Dextrose Water Hydrodissection for Carpal Tunnel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Study Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250714R
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome; Dextrose; Carpal Tunnel Release; Ultrasound; Nerve Hydrodissection Therapy
Keywords: Carpal Tunnel Syndrome; dextrose; carpal tunnel release; ultrasound; nerve hydrodissection therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- US-guided D5W perineural hydrodissection alone, group A (Active Comparator): Patients in the group A will receive 1 session of ultrasound-guided perineural injection with 5ml D5W.
  Interventions: Procedure: Active Comparator: US-guided D5W perineural hydrodissection alone, group A
- US guided partial release of the TCL with a needle + D5W injection (to TCL), group B (Active Comparator): Patients in the group B will receive 1 session of ultrasound-guided partial release of the TCL with a needle plus D5W injection to TCL.
  Interventions: Procedure: Active Comparator: US guided partial release of the TCL with a needle + D5W injection (to TCL), group B
- US-guided partial release of the TCL with D5W injection to TCL plus D5W perineural hydrodissection (Active Comparator): Patients in the group C will receive 1 session of the treatment combining group A and group B.
  Interventions: Procedure: Active Comparator: US-guided partial release of the TCL with D5W injection to TCL plus D5W perineural hydrodissection, group C

INTERVENTIONS:
Procedure: Active Comparator: US-guided D5W perineural hydrodissection alone, group A — Patients in the group A will receive 1 session of ultrasound-guided perineural injection with 5ml D5W.
  Arms: US-guided D5W perineural hydrodissection alone, group A
Procedure: Active Comparator: US guided partial release of the TCL with a needle + D5W injection (to TCL), group B — Patients in the group B will receive 1 session of ultrasound-guided partial release of the TCL with a needle plus D5W injection to TCL.
  Arms: US guided partial release of the TCL with a needle + D5W injection (to TCL), group B
Procedure: Active Comparator: US-guided partial release of the TCL with D5W injection to TCL plus D5W perineural hydrodissection, group C — Patients in the group C will receive 1 session of the treatment combining group A and group B. Hydrodissection of the median nerve will be performed before TCL release.
  Arms: US-guided partial release of the TCL with D5W injection to TCL plus D5W perineural hydrodissection

SUMMARY:
Carpal tunnel syndrome (CTS) is a common musculoskeletal disorder, which is caused by compression of the median nerve as it travels through the wrist. There are several treatments for CTS, including conservative and surgical options. Though local corticosteroid injection has been considered more effective than physical therapy for treatment of CTS and has significant short-term benefits, long term benefits are not evidenced. Several studies in recent years reported significantly superior longer-term benefit of D5W and PRP compared with corticosteroid injections and other conservative managements. In addition, percutaneous release of the transverse carpal ligament (TCL) was developed to treat CTS in recent years. Because the effectiveness of the recently developed techniques in treating CTS has not been well established, the investigators aim to investigate whether combining US-guided partial release of the transverse carpal ligament with a needle plus D5W hydrodissection is more beneficial for CTS comparing to either treatment alone.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common musculoskeletal disorder, which is caused by compression of the median nerve as it travels through the wrist. The prevalence of CTS ranges from 3% to 7.43%, and it carries a significant economic burden, influencing the number of workdays lost. Risk factors for CTS include occupations that need repetitive hand movements, female gender, age, pregnancy, obesity, diabetes, and specific anatomical and physiological traits. The symptoms and signs of CTS include tingling, numbness, nocturnal paresthesia, and pain in the median nerve distribution, whereas thenar atrophy and weakness of grasping manifest in the late stages. The widely-accepted pathophysiology includes increased pressure in the carpal tunnel, median nerve microcirculation injury, synovial tissue hypertrophy, and connective tissue compression of the median nerve. The interactions of mechanisms can lead to venous outflow obstruction, edema, and then ischemia and nerve injury ultimately. The diagnosis of CTS is made via the patient's history and physical examination, and electrodiagnostic tests may be done to differentiate among diagnoses. In recent years ultrasonographic image study of the median nerve can be applied in the evaluation and/or diagnosis of CTS. There are several treatments for CTS, including conservative and surgical options. For mild to moderate CTS, non-surgical treatments such as splinting, physical therapy, ultrasound (US)-guided corticosteroid injection, oral medications, and manual therapies are recommended. Although a systemic review showed that surgical approach yield better midterm and long term outcomes than conservative managements, there are some complications of open carpal tunnel release, including neuroma of the palmar cutaneous branch of the median nerve, infection, hypertrophic scars, postoperative pain, and persistent or recurrent symptoms. Therefore, surgical treatment is recommended only after 7 conservative management failure, or for more severe CTS.

Though local corticosteroid injection has been considered more effective than physical therapy for treatment of CTS and has significant short term benefits, long term benefits are not evidenced. In the recent decade, ultrasound guided regenerative medicine was developed to treat CTS, among which five percent dextrose in water (D5W) and platelet-rich plasma (PRP) are two commonly used injectates. Several studies in recent years reported significantly superior longer-term benefit of D5W and PRP compared with corticosteroid injections and other conservative managements. The mechanism of regenerative medicine for CTS can be divided into pharmacological and mechanical effects. The pharmacological effect includes initiating tissue proliferation in the absence of inflammation, whereas the mechanical effect can be refer to hydrodissection. In addition, percutaneous release of the transverse carpal ligament (TCL) was developed to treat CTS in recent years.

Acupotomy, using a needle-knife derived from traditional Chinese medicine to release TCL and promote local blood circulation, is a safe and effective option when performed via ultrasound guidance. Other than using a needle-knife, partial release of TCL with a needle is another choice. In a prospective study in 2022, ultrasound guided partial release of TCL using an 18-G needle was done in patients with CTS, and the result revealed that 86.2% wrists showed successful treatment outcomes at 6 months after intervention. Another cohort study in 2024 showed that treating severe CTS with ultrasound-guided partial release of TCL using a 21-G curved needle resulted in improved outcomes at the 6-week follow-up. Because the effectiveness of the recently developed techniques in treating CTS has not been well established, the investigators aim to investigate whether combining US-guided partial release of the transverse carpal ligament with a needle plus D5W hydrodissection is more beneficial for CTS comparing to either treatment alone. The investigators hypothesize that adding percutaneous release of the TCL to D5W hydrodissection could bring more therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 to 80 years old
* diagnosed with CTS on the basis of clinical condition and an electrophysiological analysis
* the NRS of pain or paresthesia≧3
* with symptoms lasting for a minimum of 3 months.

Exclusion Criteria:

* history of polyneuropathy, thoracic outlet syndrome, brachial plexopathy, or inflammatory arthropathy
* onset of CTS during pregnancy, hypothyroidism, or systemic infection
* previous corticosteroid injection or wrist surgery for CTS
* hypersensitivity to dextrose injection
* the anatomic structure of the wrist is not suitable for needle release of TCL.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a widely applied patient-reported tool for assessing the severity of carpal tunnel syndrome. This instrument consists of two sections: the Symptom Severity Scale (SSS), comprising 11 questions, and the Functional Status Scale (FSS), containing 8 items. Both scales use a 1 to 5 rating system. The minimum score is 19, and maximum value is 95. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  Pain or paresthesia severity will be assessed using the NRS, ranging from 0 (no pain and no paresthesia) to 10 (the worst imaginable pain or abnormal sensation).
Cross-sectional area (CSA) | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  Cross-sectional area (CSA) of the median nerve: The CSA of the median nerve will be assessed with an freehand tracing tool at the level of the scaphoid-pisiform, a site where median nerve swelling provides a consistent parameter for post-injection monitoring. Each measurement will be performed three times, and the average value is used for subsequent analysis.
Electrophysiological measurement | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  Assessment of the antidromic sensory nerve conduction velocity (SNCV) and distal motor latency (DML) of the median nerve will be conducted following established protocols. For SNCV measurement, surface electrodes is placed over the proximal and distal interphalangeal joints of the second digit, serving as the active and reference electrodes, respectively, with electrical stimulation applied 14 cm proximal to the active electrode along the course of the median nerve. For DML evaluation, the active electrode is positioned over the abductor pollicis brevis muscle, while the reference electrode is placed at the distal muscle-tendon junction; the median nerve is stimulated 8 cm proximal to the active electrode.
Tip pinch strength | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  Tip pinch strength, defined as the contact between the thumb pulp and index finger pulp, was assessed using a calibrated B&L pinch meter (B&L Engineering). Participants were seated with the shoulder adducted and in a neutral rotational position, the elbow flexed at 90 degrees, and the forearm and wrist placed in pronation to facilitate the measurement. Each subject performed three maximum-effort trials, with a one-minute rest period between each trial to prevent muscle fatigue. The mean value from the three trials was calculated for further analysis.
Self-assessment of the treatment effect | baseline (before injection) and at follow-up intervals of 1, 3, and 6 months after the injection.
  Self-assessment of the treatment effect All participants provided self reported evaluations of the treatment effect at 1, 3, and 6 months following the injection, using a 5-point Likert scale: much improved, improved, no change, worse, or much worse. Responses of "much improved" or "improved" were classified as indicating a positive treatment outcome. (This item is not evaluated at baseline.).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan